CLINICAL TRIAL: NCT05196100
Title: Acceptability of an Interim Socket System in the Immediate Rehabilitation of People With a tranSTibial Amputation (ASSIST): A Pilot Study
Brief Title: Acceptability of an Interim Socket System
Acronym: ASSIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government); University Hospitals Dorset NHS Foundation Trust (Other Government); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS149-291816-NV
Record Dates: First submitted 2021-12-06; First posted 2022-01-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Amputation
Keywords: transtibial; below-knee; prosthesis; socket; residual limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Confidence socket (Experimental): Participants to receive a confidence socket system
  Interventions: Device: Amparo confidence socket

INTERVENTIONS:
Device: Amparo confidence socket — Confidence socket involves thermoplastic material being moulded onto the patient's residual limb and a socket is produced in a single session. The socket can be remoulded to adjust to changes in residual limb volume.

SUMMARY:
This study will explore the acceptability of an interim socket system to new patients with a below-knee amputation and also to NHS healthcare providers.

DETAILED DESCRIPTION:
After a transtibial amputation, post-operative swelling, followed by muscle wasting, can lead to residual limb volume changes during the first 12 months. Managing this volume change often involves many socket modifications and/or replacement sockets. These multiple re-casts can be burdensome for the patient and delay recovery as patients are unable to mobilise and progress in an ill-fitting socket, leading to increased health resource use and costs.

An alternative technology exists involving an interim (aka confidence) socket whereby thermoplastic material is moulded onto the patient's residual limb and a socket is produced in a single session. This material can then be heated and remoulded quickly and comfortably, so that the patient accommodates to a single socket that can be adjusted as required to volume changes.

The confidence socket system could make the casting and prosthetic fitting process more efficient and cost-effective and improve the speed of delivery of the interim prosthesis. Thus a patient could start gait re-training with their confidence socket earlier compared to the standard treatment of fitting a laminate or polypropylene socket.

The aim of this pilot study is to assess the acceptability of the confidence socket to NHS healthcare providers and their patients, during an initial 3-month prosthetic fitting period.

Amputee participants will be recruited from 2 NHS sites. They will receive standard pre-prosthetic physiotherapy treatment until their primary MDT appointment, when they will be cast for their first prosthesis using the confidence socket which will replace standard care with the usual socket. Prescription of prosthetic foot components will continue as per usual care. Once the confidence socket is complete the patient will begin treatment according to usual physiotherapy rehabilitation. Amputee participants will be interviewed about their experience of receiving treatment with the confidence socket.

Healthcare providers delivering the treatment will also be interviewed about their acceptability of the confidence socket within the NHS pathways.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* New transtibial amputation within the last 6 months
* Deemed ready to cast for a prosthesis by the clinical team as per usual care at the prosthetic centre
* Able to understand written English and provide informed consent

Exclusion Criteria:

* Participants under the age of 18
* Participants with an ankle disarticulation, Knee disarticulation or transfemoral amputation
* Body mass > 125 kg with a distal circumference of 23-34 cm (small socket)
* Body mass > 150 kg with a distal circumference of 30-45 cm (large socket)
* Residual limb longer than 27 cm
* Severe upper limb dysfunction (due to strength requirements to don the liner)
* Severe visual requirements (that would restrict the person's ability to monitor their residual limb)
* Contraindication to be fit for a prosthetic socket
* Recent cerebrovascular event (i.e., stroke, haemorrhage, brain injury)
* Disease affecting their memory
* Unwilling to trial the confidence socket system
* Unable to tolerate wearing a prosthetic liner due to excess sweating/ allergic reaction or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-11-28 (Estimated); Study Completion 2024-11-28 (Estimated)

PRIMARY OUTCOMES:
Change in Socket comfort score | Up to 6 months
  Patient-reported socket comfort

SECONDARY OUTCOMES:
Change in EQ-5D-5L | Up to 6 months
  Health related quality of life
Change in Locomotor Capabilities Index (LCI-5) | Up to 6 months
  LCI-5 with prosthesis
Change in Activities Balance Confidence-UK (ABC-UK) | Up to 6 months
  Balance confidence
Change in L-test | Up to 6 months
  Functional timed up and go L-test

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth
  - Portsmouth Hospitals University NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No